CLINICAL TRIAL: NCT06250881
Title: Analysis of Ocular Complications of AIDS Patients in Ophthalmic Consultation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20231119
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-11

CONDITIONS: Ocular Complications in AIDS Patients, Such as Fundus Opportunistic Infections, Microangiopathy, and Uveitis
Keywords: Ocular complications of AIDS
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- without ocular complication: The normal group was compared with the pathological group
- fundus opportunistic infections: AIDS patients are prone to opportunistic fundus infection, which show a characteristic changes in fundus photography. It was designed to describe the characteristics of this group of patients.
- Microvascular disease: Microvascular disease is an early characteristic of fundus changes in AIDS patients, with characteristic changes in fundus photography.
- uveitis: The uveitis patients in this study were mainly caused by treponema pallidum infection.

SUMMARY:
Through a cross-sectional descriptive analysis of ophthalmic consultation of AIDS patients in the past 3 years, the basic characteristics of patients were described according to whether there was fundus change, and the clinical characteristics and risk factors of CMVR patients with or without RD were compared.

DETAILED DESCRIPTION:
Patients were divided into normal group, opportunistic infection group, microangiopathopathy group and uveitis group according to the presence of fundus lesions and the types of fundus lesions. The basic information and characteristics of patients in different groups were described. The factors that may be related to ocular fundus disease of AIDS patients were found by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* AIDS inpatient undergoing ophthalmic consultation

Exclusion Criteria:

* Non-hiv infected patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV/AIDS patients hospitalized in the infection department at ZhongNan Hospital with ophthalmic consultation during November 19th, 2019 to June 9th ,2023 were included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-28 (Estimated)

PRIMARY OUTCOMES:
fundus photo changes | The classification was based on a review of the fundus examination of the patient at the time of the 1 day visit
  Early changes(microangiopathy) appear as small, white, scattered retinal infiltrations. And the typical change of CMVR is full-layer, cheesy retinal necrosis with extensive retinal bleeding in the distal region.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yen M, Chen J, Ausayakhun S, Kunavisarut P, Vichitvejpaisal P, Ausayakhun S, Jirawison C, Shantha J, Holland GN, Heiden D, Margolis TP, Keenan JD. Retinal detachment associated with AIDS-related cytomegalovirus retinitis: risk factors in a resource-limited setting. Am J Ophthalmol. 2015 Jan;159(1):185-92. doi: 10.1016/j.ajo.2014.10.014. Epub 2014 Oct 22. PMID 25448999
- [Result] De Cock KM, Jaffe HW, Curran JW. Reflections on 40 Years of AIDS. Emerg Infect Dis. 2021 Jun;27(6):1553-1560. doi: 10.3201/eid2706.210284. PMID 34013858
- [Result] Landovitz RJ, Scott H, Deeks SG. Prevention, treatment and cure of HIV infection. Nat Rev Microbiol. 2023 Oct;21(10):657-670. doi: 10.1038/s41579-023-00914-1. Epub 2023 Jun 21. PMID 37344551
- [Result] Bekker LG, Beyrer C, Mgodi N, Lewin SR, Delany-Moretlwe S, Taiwo B, Masters MC, Lazarus JV. HIV infection. Nat Rev Dis Primers. 2023 Aug 17;9(1):42. doi: 10.1038/s41572-023-00452-3. PMID 37591865
- [Result] Cohn LB, Chomont N, Deeks SG. The Biology of the HIV-1 Latent Reservoir and Implications for Cure Strategies. Cell Host Microbe. 2020 Apr 8;27(4):519-530. doi: 10.1016/j.chom.2020.03.014. PMID 32272077